CLINICAL TRIAL: NCT06384183
Title: Kerecis Real-World Fish Skin Graft Registry - "ISACOD"
Brief Title: Kerecis Real-World Fish Skin Graft Registry
Acronym: ISACOD
Status: Enrolling by invitation | Type: Observational
Sponsor: Kerecis Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: KS-1000
Record Dates: First submitted 2024-04-22; First posted 2024-04-25 (Actual); Last update posted 2024-12-30 (Actual); Status verified 2024-08

CONDITIONS: Wounds; Pressure Ulcer; Diabetic Foot Ulcer; Venous Leg Ulcer; Surgical Wound; Soft Tissue Reinforcement
MeSH Terms: conditions — Wounds and Injuries; Pressure Ulcer; Diabetic Foot; Varicose Ulcer; Surgical Wound

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Observational Group: This observational (i.e., non-interventional), post-market, real-world, Registry was designed to collect, analyze, and identify relevant safety and performance outcomes for "all comers" using Kerecis devices in routine medical practice within a wide variety of United States (US) medical practice settings.
  Interventions: Device: Kerecis Fish Skin Graft

INTERVENTIONS:
Device: Kerecis Fish Skin Graft — Patients already treated with a Kerecis device

SUMMARY:
Multi-center, observational (i.e., non-interventional), open-label, real-world Registry on the Use of Kerecis Devices

DETAILED DESCRIPTION:
This observational (i.e., non-interventional), post-market, real-world, Registry was designed to collect, analyze, and identify relevant safety and performance outcomes for "all comers" using Kerecis devices in routine medical practice within a wide variety of United States (US) medical practice settings. These clinical data will be used at Kerecis for many purposes, which include, but are not limited to, device safety and performance evaluation as part of routine patient care and post-market clinical follow-up data commitments to regulatory authorities around the world.

ELIGIBILITY:
Inclusion Criteria:

* Provided informed consent
* Has at least one target wound treated with a Kerecis device according to physician medical judgement within one calendar month prior to the registry enrollment date

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Investigators will only enter previously collected clinical data from patients (all ages, demographics, and any health status) who meet all inclusion criteria and no exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2024-08-07 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Fish Skin Graft Device Related failure | 12 months
  Proportion of patients with Kerecis FSG device-related failure for any reason (e.g., resulting in non-absorption or device removal)
Fish Skin Graft Device related allergy | 12 months
  Proportion of patients with Kerecis FSG device-related allergy, hypersensitivity and/or autoimmune reaction (with or without documented auto-antibody development)
Target Wound Infection | 12 months
  Proportion of patients who develop target wound infection

SECONDARY OUTCOMES:
Complete Wound Healing | 12 months
  The Time in weeks to complete healing
Complete Wound Closure | 12 months
  Proportion of participants who experience complete wound closure

CONTACTS AND LOCATIONS:
Overall Officials: Anne Swearingen, Principal Investigator — Kerecis Ltd.
Locations (6):
- United States (6):
  - MCR Health, Sarasota, Florida
  - University Park, Sarasota, Florida
  - Cone Health Ortho Care Greensboro, Greensboro, North Carolina
  - Feet First Institute of Beavercreek, Beavercreek, Ohio
  - ABC Podiatry, Columbus, Ohio
  - South Texas Skin Cancer Center, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: Undecided
To be determined